CLINICAL TRIAL: NCT00011973
Title: A Phase Two Study Of Fenretinide In Renal Cell Cancer
Brief Title: Chemotherapy in Treating Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068465; U01CA062487 (NIH); P30CA022453 (NIH); WSU-C-2232; NCI-WSU-910
Record Dates: First submitted 2001-03-03; First posted 2003-08-08 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Fenretinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fenretinide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of fenretinide in treating patients who have advanced kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with advanced renal cell carcinoma treated with fenretinide.
* Determine progression-free and overall survival of this patient population treated with this drug.
* Determine the quantitative and qualitative toxic effects of this drug in these patients.

OUTLINE: Patients receive oral fenretinide twice a day for 7 days. Courses repeat every 21 days in the absence of unacceptable toxicity or disease progression.

PROJECTED ACCRUAL: Approximately 18-35 patients will be accrued for this study within 9-21 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed locally advanced unresectable, locally recurrent, or metastatic renal cell carcinoma
* Measurable disease

  * At least 20 mm with conventional techniques OR
  * At least 10 mm with spiral CT scan
* No nonmeasurable disease only including:

  * Bone lesions
  * Leptomeningeal disease
  * Ascites
  * Pleural/pericardial effusion
  * Lymphangitis cutis/pulmonis
  * Abdominal masses not confirmed and followed by imaging techniques
  * Cystic lesions
* No known brain metastases

  * History of brain metastases that have been resected and/or irradiated with subsequent normal brain CT scan allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy:

* More than 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 2 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior malignancy within the past 2 years except nonmelanoma skin cancer or carcinoma in situ of any site
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to fenretinide
* No other concurrent uncontrolled illness (e.g., ongoing or active infection)
* No concurrent psychiatric illness or social situation that would preclude study
* History of HIV allowed if no active infection or history of retinitis
* No history of retinal disease, night blindness, or difficulty seeing in the dark

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior biologic therapy allowed

Chemotherapy:

* No more than 1 prior chemotherapy regimen

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics

Other:

* Recovered from prior therapy
* No prior systemic retinoid therapy
* No concurrent antioxidants (e.g., ascorbic acid or vitamin E)
* No other concurrent therapy for renal cell carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulka N. Vaishampayan, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (4):
- United States (4):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Vaishampayan U, Heilbrun LK, Parchment RE, Jain V, Zwiebel J, Boinpally RR, LoRusso P, Hussain M. Phase II trial of fenretinide in advanced renal carcinoma. Invest New Drugs. 2005 Mar;23(2):179-85. doi: 10.1007/s10637-005-5864-7. PMID 15744595